CLINICAL TRIAL: NCT06847425
Title: Sphenopalatine Ganglion Block with Bupivacaine and Its Effect on Pain After Functional Endoscopic Sinus Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FMASU MS221/2024
Record Dates: First submitted 2025-02-21; First posted 2025-02-26 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-01

CONDITIONS: Anaesthesia

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (control group) (n= 35 ) (Active Comparator): 1.5 ml of normal saline was injected in the greater palatine foramen
  Interventions: Procedure: Sphenopalatine Ganglion Block trans oral approach saline injection
- Group B (Bupivacaine group) (n= 35) (Active Comparator): 1.5 ml of Bupivacaine was injected in the greater palatine foramen.
  Interventions: Procedure: Sphenopalatine ganglion block trans oral approach bupivacaine injection

INTERVENTIONS:
Procedure: Sphenopalatine Ganglion Block trans oral approach saline injection — The sphenopalatine block will be done by the end of the operation using a trans-oral approach at the greater palatine foramen with the help of a Macintosh blade number 3 for good visualization of the hard and soft palate using a 25 Gauge 1.5 inch needle curved at 45 degrees 25 mm from the tip and filled with 1.5 ml of normal saline. The greater palatine foramen is located posteromedial to the third maxillary molar and anteromedial to the pterygoid hamulus and maxillary tuberosity. The foramen will be identified by digital palpation, and the needle will be inserted until reaching the bone then redirected slightly until the foramen is localized and the needle easily gets in the greater palatine canal. aspiration will be done to ensure that no blood vessels are punctured, and the solution will be injected.
  Arms: Group A (control group) (n= 35 )
Procedure: Sphenopalatine ganglion block trans oral approach bupivacaine injection — The sphenopalatine block will be done by the end of the operation using a trans-oral approach at the greater palatine foramen with the help of a Macintosh blade number 3 for good visualization of the hard and soft palate using a 25 Gauge 1.5 inch needle curved at 45 degrees 25 mm from the tip and filled with 1.5 ml of bupivacaine. The greater palatine foramen is located posteromedial to the third maxillary molar and anteromedial to the pterygoid hamulus and maxillary tuberosity. The foramen will be identified by digital palpation, and the needle will be inserted until reaching the bone then redirected slightly until the foramen is localized and the needle easily gets in the greater palatine canal. aspiration will be done to ensure that no blood vessels are punctured, and the solution will be injected.
  Arms: Group B (Bupivacaine group) (n= 35)

SUMMARY:
Functional endoscopic sinus surgery (FESS) is a minimally invasive procedure that is used in many inflammatory and infectious sinus diseases. Acute postoperative pain can lead to adverse consequences and good postoperative treatment of pain is essential. There is no agreement on a single protocol to treat pain after endoscopic sinus surgeries, and the usually used analgesics have some side effects that hinder their use. Current evidence is insufficient for routine clinical use of the sphenopalatine ganglion block for Functional endoscopic sinus surgery and the efficacy of sphenopalatine ganglion block for pain control after functional endoscopic sinus surgery remains controversial. This study aims to explore the influence of sphenopalatine ganglion block on pain intensity after functional endoscopic sinus surgery by comparing two groups, a group receiving the block with Bupivacaine injection, versus saline injection in the other group.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18 years - 80 years.
2. ASA I and ASA II patients.
3. Consented to participate in the research.

Exclusion Criteria:

1. Pregnant and breastfeeding females.
2. History of allergy to bupivacaine or other local anaesthetics.
3. Patients with uncontrolled hypertension, poorly controlled cardiovascular diseases, or cerebrovascular diseases.
4. Patients with pre-existing neurological conditions.
5. Patients with history of alcohol or drug abuse.
6. Patients on anticoagulation.
7. Occurrence of surgical or anaesthetic complications or change in the anaesthesia protocol.
8. Patients showing sensitivity to Bupivacaine.
9. Patients unable to understand VAS score.
10. Patients refusing to continue participating in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2024-03-20 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2024-08-30 (Actual)

PRIMARY OUTCOMES:
Mean Visual Analogue Scale (VAS) pain score over the first 24 hours postoperatively. | in the PACU, at 2, 6, 12, and 24 hours after surgery
  Postoperative pain will be assessed with a 10-cm scale visual analogue scale (VAS) (0 = no pain, 10 = worst imaginable pain)

SECONDARY OUTCOMES:
Time to first rescue analgesia | 24 hours postoperatively
  Participants with VAS score ≥4 at any point of time and complaining of pain will receive fentanyl (25-50 μg) as a rescue analgesic and the time to the first rescue analgesia will be recorded
Total requirements of rescue analgesia | 24 hours postoperatively
  Participants with VAS score ≥4 at any point of time and complaining of pain will receive fentanyl (25-50 μg) as a rescue analgesia
Number of patients receiving rescue analgesia | 24 hours postoperatively
  Participants with VAS score ≥4 at any point of time and complaining of pain will receive fentanyl (25-50 μg) as a rescue analgesic.
Incidence and severity of adverse effects and complications | 24 hours postoperatively
  Incidence and severity of adverse effects and complications such as nausea and vomiting (PONV), headache, visual disturbances, sore throat and swallowing difficulty during the first 24 hours postoperatively

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Egypt